CLINICAL TRIAL: NCT04707430
Title: The Effect of Progesterone Levels on the 3rd and 5th Days After Insemination on Pregnancy
Brief Title: The Effect of Progesterone Levels on Pregnancy
Status: Completed | Type: Observational
Sponsor: Sezcan Mumusoglu (Other)
Responsible Party: Sponsor-Investigator, Sezcan Mumusoglu, associated professor, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: HU1101
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Relationship of Progesterone Levels and Pregnancy
Keywords: intrauterine insemination; progesterone; pregnancy; gonadotropins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood progesterone test — progesterone levels on blood sample

SUMMARY:
The aim of this study is to investigate the effect of progesterone levels on pregnancy occurrence on the 3rd and 5th days after insemination.

DETAILED DESCRIPTION:
Ovarian stimulation with gonadotropins is a frequently used method in patients with unexplained infertility undergoing intrauterine insemination.

Pregnancy and live birth rates after ovarian stimulation; The number of follicles in ovulatory size and responsive to ovarian stimulation is affected by many factors such as the age of the woman and the duration of infertility. Progesterone production in the luteal phase is necessary to achieve successful treatment results by increasing the receptivity of the endometrium in the secretory phase.

In assisted reproductive techniques, exogenous progesterone support in the luteal phase is a routinely used method due to higher pregnancy rates, but there is no consensus with the use of progesterone in IUI applications. In a recent meta-analysis, a positive relationship was found between gonadotropins and progesterone support when ovulation induction and intrauterine insemination were performed, while this relationship was not found with clomiphene citrate, and although letrozole and gonadotropin were used together, no significant statistics were found.

The relationship between luteal phase hormone dynamics and pregnancy outcomes in IUI is not fully understood. Although luteal phase failure is mentioned, there is no accepted definition of luteal phase failure worldwide. In one study, progesterone concentrations in the midluteal phase and pregnancy outcomes were investigated in 188 IUI cycles, predicting that low levels could predict treatment failure. In another study, a positive relationship was found between luteal phase progesterone levels and clinical pregnancy outcomes.However, the relationship between blood progesterone levels and pregnancy rates in a small number of IUI cycles has been investigated in the literature. Considering all these studies, there is no Level 1 evidence regarding the benefit of providing progesterone support in groups where the progesterone level is below a certain threshold value. In this study, we aimed to investigate the relationship between gestational outcomes by looking at progesterone values on the 3rd and 5th days after IUI in patients who were decided to be treated with IUI. By looking at these progesterone levels, we aimed to determine a threshold value for the ideal level of progesterone in the luteal phase and to be a guide in terms of possible results and methods of shaping the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been decided for intrauterine insemination
* Patients under the age of 40
* Patients with a BMI of less than 40 kg / m2
* Cycles triggered by rhCG
* Those who have a signed and dated informed consent document that they have been informed about the study and that their consent has been obtained

Exclusion Criteria:

* Patients over the age of 40
* Patients with BMI over 40 kg / m2

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients admitted to Hacettepe Hospital and scheduled for insemination
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The progesterone level | up to 12 months
  the effect of progesterone levels 3rd and 5th day after insemination on ongoing pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Bozdag, Prof., Study Chair — Hacettepe University; Galip Serdar Gunalp, Prof., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)